CLINICAL TRIAL: NCT06811961
Title: Effects of Exercise on Edema, Pain, Exercise Capacity, Lower Extremity Muscle Strength and Function in Patients with Lipedema
Brief Title: Effects of Exercise in Patients with Lipedema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilke Keser (Other)
Responsible Party: Sponsor-Investigator, Ilke Keser, Prof. Dr., Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ElifSakizliLipedema
Record Dates: First submitted 2025-01-26; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Lipedema
Keywords: lipedema; exercise; function
MeSH Terms: conditions — Lipedema; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Patients with lipedema will perform group exercises consisting of warm-up, loading and cool-down periods of 40-50 minutes, 2 days a week for 6 weeks, and strengthening exercises applied to the muscles around the hips and knee extensors with elastic resistance bands, determined according to the effort level perceived by the patient, 3 sets of 10 repetitions, 2 days a week for 6 weeks.
  Interventions: Behavioral: Exercise
- Control group (Other): The control group will be given recommendations regarding lipedema and physical activity level.
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Exercise — Patients with lipedema will perform group exercises consisting of warm-up, loading and cool-down periods of 40-50 minutes, 2 days a week for 6 weeks, and strengthening exercises applied to the muscles around the hips and knee extensors with elastic resistance bands, determined according to the effort level perceived by the patient, 3 sets of 10 repetitions, 2 days a week for 6 weeks.
  Arms: Exercise group
Behavioral: Physical activity — The control group will be given recommendations regarding lipedema and physical activity level.
  Arms: Control group

SUMMARY:
Lipedema is a chronic progressive disease characterized by symmetrical, disproportionate swelling of subcutaneous adipose tissue, which is common in women and mostly seen in the lower extremities and to a lesser extent in the upper extremities. Healthy lifestyle approaches including exercise treatments are very important for lipedema patients in order to prevent disease progression. The aim of this study is to investigate the effects of exercise on edema, pain, exercise capacity, lower extremity muscle strength and function in lipedema patients. Sociodemographic information of the patients, body composition with Tanita InnerScan BC-601-CG device, clinical information regarding lipedema, type and stage of lipedema, inspection, palpation findings will be recorded. Local tissue water percentage will be assessed using Moisturemeter-d compact (MMDc, Delfin Technologies, Kuopio, Finland) device, circumference measurement using tape, pain intensity with Visual Analog Scale, pain threshold with Baseline brand digital algometer device. Muscle strength will be assessed using K-Force hand dynamometer. Functional exercise capacity will be assessed with the 6-minute walk test (6MWT), and lower extremity dysfunction with the lower extremity functional scale. After the assessments are made, the patients will be randomly divided into 2 groups. The patients in the study group will perform group exercises consisting of warm-up, loading and cool-down periods of 40-50 minutes, 2 days a week for 6 weeks, and strengthening exercises applied to the hip muscles and knee extensors with elastic resistance bands, which are decided according to the level of effort perceived by the patient, 3 sets of 10 repetitions, 2 days a week for 6 weeks. The same assessments will be applied to the patients again at the end of the exercise program. The control group will be re-evaluated after 6 weeks with suggestions regarding lipedema and physical activity level, and the obtained data will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Lipedema,
* Patients with Lipedema stage 1,2 and 3

Exclusion Criteria:

* Individuals with cardiopulmonary, rheumatic or neurological diagnoses that have symptoms severe enough to prevent participation in exercise,
* History of cancer, surgery or trauma that may affect the circulatory system,
* History of liposuction or orthopedic surgery within the last year,
* Individuals who cannot mobilize independently.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
Local tissue water percentage | 6 weeks
  Local tissue water percentage will be measured with the Moisturemeter-d compact (MMDc, Delfin Technologies, Kuopio, Finland) device. This device calculates the percentage of water under the skin by touching the reference points from the skin surface. 3 measurements will be made for each reference point and the average of these measurements will be recorded. The reference points were determined as the medial of 35 cm above the heel (calf) on both legs, the medial of 3 cm proximal to the patella (medial knee) and the lateral of 20 cm above the line drawn from 3 cm proximal to the patella to the SIAS (lateral hip).
edema | 6 weeks
  For the lower extremity, the circumference will be measured at 4 cm intervals starting from the lateral malleolus to the highest point that can be reached on the inner thigh. The circumference measurement is performed while the patient is lying on his back. The results are recorded in cm and the volume calculation will be made according to the Khunke disk method.
Pain severity | 6 weeks
  The leg pain due to lipedema will be recorded in cm with the Visual Analog Scale (VAS) according to the patient's statement.
Pain Threshold | 6 weeks
  A Baseline brand digital algometer device will be used to assess the pain threshold. A 1 cm2 probe will be used for measurements. Before the measurement process, the midpoint of the quadriceps and tibia will be marked. The measurement will be repeated three times at 5-second intervals and the average values will be recorded in kg. The algometer will be placed at a right angle to each point, the participants will be asked to report the presence of pain by saying "yes" and the value on the device will be recorded as the pain threshold when they first feel pain at the point of touch. There will be a 5-second break between measurements.
Lower extremity muscle strength | 6 weeks
  Muscle strength measurements will be made with K-Force hand dynamometer. Quadriceps Femoris and hip flexors muscle strength will be measured in sitting position and hip abductors muscle strength will be measured in side-lying position. During the measurements, patients will be asked to perform maximum isometric contraction for 5 seconds. Muscle strength measurements will be repeated 3 times on the right and left sides separately and maximum value will be recorded in kg.
Lower extremity muscle endurance | 6 weeks
  Lower extremity muscle endurance measurement will be evaluated with a 30-second sit-to-stand test. The patient will be asked to stand up and sit down from a back-supported chair with their arms crossed on both shoulders for 30 seconds. Sitting down and standing less than 10 times in 30 seconds indicates a loss of lower extremity strength.
functional exercise capacity | 6 weeks
  Exercise capacity will be evaluated with a 6-minute walking test. The distance covered will be recorded and interpreted as normal values. Heart rate and oxygen saturation will be measured with a portable pulse oximeter before and after the test; blood pressure will be measured with a device that automatically measures (Omron-Hem 710 Int, USA). Dyspnea and fatigue levels will be evaluated with the Modified Borg Scale (MBS) at the beginning and end of the test. The Modified Borg Scale is a scale that evaluates fatigue and shortness of breath between 0-10.
lower extremity function | 6 weeks
  The lower extremity functional scale is a questionnaire consisting of 20 items developed to evaluate the lower extremity functions of patients. There are 5 options from 0 to 4 for each question (0: Extreme difficulty or inability to perform the activity, 1: Quite a bit of difficulty, 2: Moderate difficulty, 3: Some difficulty, 4: No difficulty at all). The total score varies between 0-80 and higher scores indicate better functional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Health Sciences, Ankara, Emek, Turkey (Türkiye)

REFERENCES:
- [Derived] Sakizli Erdal E, Ergin C, Haspolat M, Erturk B, Keser I. Effects of multimodal exercise program on edema, pain, exercise capacity, lower extremity muscle strength and function in patients with lipedema. Phlebology. 2026 Feb;41(1):47-57. doi: 10.1177/02683555251343148. Epub 2025 May 15. PMID 40372970